CLINICAL TRIAL: NCT03897764
Title: A Novel Analgesic Method for Postoperative Pain Relief After Cesarean Section: Intraoperative Superior Hypogastric Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Berna Haliloglu Peker, Prof. Dr. Berna Haliloglu Peker, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101/5.5.2017
Record Dates: First submitted 2019-03-23; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Postoperative Pain
Keywords: cesarean section; postoperative pain; superior hypogastric block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: prospective double-blinded randomized placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients were randomly allocated in two groups. The allocation sequence was generated by a random number table, and group allocation was concealed in sealed, opaque envelopes that were not opened until operation. During the operation the envelope was opened by a nurse outside the operating theatre. The nurse prepared a blind syringe with the study drug, which was then transferred to a sterile bowl in the operating room and injected. Both bupivacaine and saline are colourless and not possible to identify the solution by its visual appearance, or by smell. The envelope was then sealed again and not opened until the study was concluded. The patients, anesthesiologists, and nurses providing postoperative care were blinded to group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Superior Hypogastric Block group (Experimental): The group which superior hypogastric block performed intraoperatively
  Interventions: Procedure: Intraoperative superior hypogastric plexus block
- placebo controlled group (Placebo Comparator): The group which placebo used
  Interventions: Procedure: Intraoperative superior hypogastric plexus block

INTERVENTIONS:
Procedure: Intraoperative superior hypogastric plexus block — SHP is situated anterior to L5-S1 vertebral bodies, caudal to the bifurcation of the aorta. An injection of 20 ml of bupivacaine 2,5 mg/ml or saline 9 mg/ml was done retroperitoneally in the area.

SUMMARY:
Cesarean section is the most common inpatient surgical procedure in the United States with 1.3 million cesarean deliveries performed in 2015. Cesarean section frequency is increasing rapidly in worldwide, especially in middle and high income countries.

Postoperative pain is an expected outcome for patients following surgical procedures. Inadequate pain relief is still a common problem among hospitalized patients. Cesarean section ranked ninth for pain severity among 179 different surgical procedures.

Multimodal pain therapy has been suggested for postoperative pain management after cesarean delivery. The most commonly used modalities are systemic administration of opioids, either by intramuscular injection or IV by patient-controlled analgesia, and neuraxial injection of opioid as part of a regional anesthetic for cesarean delivery. These techniques have specific advantages and disadvantages.

Superior hypogastric plexus blockade (SHB) has been shown an effective method for pain relıef after gynecologic procedures, it has been shown that SHP can be easily performed intraoperatively during hysterectomy procedure In this study, we aimed to investigate the efficacy of SHB performed intraoperatively for postoperative pain relief after cesarean section. To our knowledge, this is the first study to use SHB intraoperatively for pain relief after cesarean section in the literature.

DETAILED DESCRIPTION:
Cesarean section is a life-saving surgical operation performed during pregnancy and labor. It is the most common inpatient surgical procedure in the United States with 1.3 million cesarean deliveries performed in 2015. Cesarean section frequency is increasing rapidly in worldwide, especially in middle and high income countries.

Postoperative pain is an expected outcome for patients following surgical procedures. Inadequate pain relief is still a common problem among hospitalized patients. A number of surveys report that 30%-70% of surgical patients experience moderate to severe pain (Breivik) At least 10.9% of women experience severe pain within 24 h after cesarean section. An analysis of 50523 patients from 105 hospitals questioning pain intensity on the first postoperative day revealed that cesarean section ranked ninth for pain severity among 179 different surgical procedures.

In this regard, multimodal pain therapy has been suggested for postoperative pain management after cesarean delivery. It requires the use of a combination of drugs with different mechanisms of action, and aims at achieving optimal analgesia through additive or synergistic drug action with small doses of opiates and decreased side effects. The most commonly used modalities are systemic administration of opioids, either by intramuscular injection or IV by patient-controlled analgesia, and neuraxial injection of opioid as part of a regional anesthetic for cesarean delivery. These techniques have specific advantages and disadvantages.

Recently, superior hypogastric plexus blockade (SHB) has been shown an effective method for pain relıef after gynecologic procedures, i.e. hysterectomy (kaynak). The superior hypogastric plexus (SHP) is a retroperitoneal structure located bilaterally at the level of the lower third of the fifth lumbar vertebral body and upper third of the first sacral vertebral body at the sacral promontory in which it is most accessible to block for pelvic pain relief. Besides it can be performed either by fluoroscopy-guided, ultrasound (US)-guided, or CT-guided techniques, it has been shown that SHP can be easily performed intraoperatively during hysterectomy procedure ().

In this study, we aimed to investigate the efficacy of SHB performed intraoperatively for postoperative pain relief after cesarean section. To our knowledge, this is the first study to use SHB intraoperatively for pain relief after cesarean section in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Term singleton pregnant women between ages 18 to 40 with no previous history of cesarean section or abdominal surgery were scheduled for elective cesarean operation under general anaesthesia. Only ASA 1-2 patients were included to the study.

Exclusion Criteria:

* We excluded patients with suspected or manifest bleeding disturbances, chronic pelvic pain, allergy to NSAID's or opioids, atopia, bronchial asthma, diabetes mellitus, the presence of liver or kidney diseases, abuse of drugs or alcohol, and patients with pregnancy-induced hypertension or preeclampsia. The patients underwent emergency cesarean section were also excluded from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women scheduled for cesarean operation eligible fot he study
Enrollment: 154 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Pain scores on rest and on movement at 24 th hour after surgery | up to 24 hours
  Postoperative pain assessed by the 10 cm visual analogue scale (VAS) ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable

SECONDARY OUTCOMES:
Pain scores on rest and on movement at 2,6 and 48 th hour after surgery | Up to 48 hours
  Postoperative pain assessed by the 10 cm visual analogue scale (VAS) ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable
Opioid or NSAID requirement after surgery | Up to 48 hours
  Total opioid and NSAID requirement for postoperative pain relief after surgery were calculatedcalculated
Return of gastrointestinal function | Up to 48 hours
  First passage of flattus was noted as a sign of bowel function
Rate of nausea and vomiting | Up to 48 hours
  Rate of nausea and vomiting as a side effect of the procedure
length of surgery | Up to 1 hour
  length of cesarean section was recorded in each group

CONTACTS AND LOCATIONS:
Overall Officials: Berna Haliloglu Peker, Prof. Dr, Principal Investigator — Maltepe University Faculty of Medicine
Locations (1):
- Maltepe University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT03897764/Prot_SAP_000.pdf